CLINICAL TRIAL: NCT05714384
Title: Outcome of Calcium Silicate Sealer-based Obturation in Root Canal Retreatment: A CBCT-based Prospective Cohort Study
Brief Title: Calcium Silicate Sealer-based Obturation in Root Canal Retreatment
Status: Enrolling by invitation | Type: Observational
Sponsor: Ministry of Health, Kuwait (Other Government)
Collaborators: Kuwait Institute for Medical Specialization (Other Government)
Responsible Party: Principal Investigator, Ahmed Aldowaisan, Principal Investigator, Specialist in Endodontics, Ministry of Health, Kuwait
Other Study IDs: 2238
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Root Canal Infection; Periapical Diseases
MeSH Terms: conditions — Periapical Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CeraSeal (Calcium Silicate-based Root Canal Sealer) — A calcium silicate-based root canal sealer will be used in cases requiring root canal retreatment.

SUMMARY:
This study will evaluate the outcome of calcium silicate sealer-based obturations in root canal retreatment.

DETAILED DESCRIPTION:
Calcium silicate sealer-based obturations have shown promising performance in primary root canal treatments, but there is a lack of prospective studies evaluating their effectiveness in secondary root canal treatments, which often involve more persistent microbial challenges. The aim of this study is to assess the clinical and radiographic outcomes of calcium silicate sealer-based obturations in root canal retreatment and to identify potential prognostic factors for healing.

Objectives:

1. To determine the success rate of calcium silicate sealer-based obturations in root canal retreatment.
2. To compare the observed outcomes with previously published retreatment studies using conventional obturation techniques.
3. To identify potential prognostic factors associated with favourable or unfavourable outcomes.

This will be a prospective cohort study conducted at Jaber Al-Ahmed Dental Center. Informed written consent will be obtained from all participants. All nonsurgical root canal retreatments will be performed by a specialist endodontist using a calcium silicate-based sealer (CeraSeal, Meta Biomed) following current evidence-based standards. Treatments will be recorded in a secure database, and all cases will be followed for a minimum of 12 months.

Clinical and radiographic records will be reviewed, and eligibility will be determined according to predefined inclusion and exclusion criteria. All patient data will be anonymized before extraction and analysis.

The primary outcome at 12 months will be the proportion of teeth classified as having a favourable outcome. This outcome will serve as the dependent variable in logistic regression models evaluating the associations between healing and potential predictors, including age, sex, tooth type, periapical status, preoperative pain, quality of the previous root filling, sinus tracts, presence of exudate, apical patency, final apical preparation size, sealer extrusion, and duration of intracanal medication. Separate univariable logistic regression models will be performed for each predictor. A multivariable logistic regression model will then be constructed to evaluate the combined effects of independent variables, with exploratory assessment of two-way interactions.

This study was designed as a single-arm prospective outcome investigation with the primary endpoint being the proportion of teeth exhibiting a favourable outcome. A precision-based approach was used to determine the required sample size. An anticipated healing rate of 80 percent was assumed based on systematic reviews (Ng et al. 2008; Sabeti et al. 2024; Martins et al. 2025) and prospective cohort studies (Ng et al. 2011; Davies et al. 2015; Nuaimi et al. 2017) that report healing rates between 77 and 87 percent for nonsurgical retreatment.

Using PASS (version 25.0.3; NCSS, LLC, Kaysville, Utah, USA) with the One Proportion - Confidence Interval procedure (two-sided 95 percent confidence level, Wilson method), a sample size of 95 teeth was required to estimate the healing proportion with a target precision of approximately ±8 percentage points. Allowing for up to 30 percent attrition, the planned enrolment was set at 136 teeth, which is expected to yield at least 95 evaluable cases. This target aligns with sample sizes used in previous prospective clinical studies on endodontically retreated teeth (Davies et al. 2015; Karaoğlan et al. 2022; Serefoglu et al. 2022).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18-65 years of age at the time of recruitment
* Participants must have a classification of I or II on the American Society of Anesthesiologists (ASA) physical status classification system
* Participants must not have known allergies to any materials used in the study
* Participants must agree to participate in the study by signing a consent form
* Participants must have good oral hygiene
* All types of permanent teeth that require root canal retreatment are included (incisors, canines, premolars & molars)
* The teeth must be restorable and have fully formed roots with no advanced periodontal disease

Exclusion Criteria:

* ASA classification of III or more
* Pregnant or breastfeeding women
* Patients who are unable to give consent
* Patients who have advanced periodontal disease or teeth with more than 5mm probing
* Teeth with incomplete root formation
* Teeth that have a poor restorative prognosis
* Teeth presenting with signs of a vertical root fracture
* Teeth with blocked or non-negotiable canals
* Teeth with broken instruments
* Teeth with iatrogenic perforations
* Teeth requiring posts or extensive prosthetic rehabilitation
* Teeth with cracks
* Teeth with internal or external root resorption
* Teeth with uncontrollable exudate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who present with symptomatic teeth and require root canal retreatment will be assessed based on inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 136 (Estimated)
Dates: Start 2023-03-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of radiographic healing with cone beam computed tomography (CBCT) scans using Estrela's PAI (periapical index) | Comparison of periapical lesion size at baseline and 12 months
  Estrela's PAI based on CBCT will be used in logistic regression models with different predictor variables.
Assessment of clinical outcome by assessing the resolution/persistence/development of clinical signs and symptoms | Comparison at baseline and 12 months
  The examiner will label the teeth as having a normal clinical outcome (absence of pain, swelling and other symptoms, no sinus tract, no loss of function) or showing signs and symptoms clinical outcome (the tooth is associated with signs and/or symptoms of infection).

CONTACTS AND LOCATIONS:
Locations (1):
- Jaber Al-Ahmed Dental Center, Janūb as Surrah, Hawalli Governate, Kuwait

IPD SHARING:
Plan to Share IPD: No
IPD will not be available to other researchers.